CLINICAL TRIAL: NCT03187067
Title: Evaluation of Impact of Lung Ultrasound (LUS) on Management of Pneumonia in Low-resource Settings
Brief Title: Pediatric Pneumonia Lung Ultrasound
Acronym: PLUS
Status: Completed | Type: Observational
Sponsor: Save the Children (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Barcelona Institute for Global Health (Other); Aga Khan University (Other)
Responsible Party: Sponsor
Other Study IDs: PLUS
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pneumonia; Acute Respiratory Infection
Keywords: pneumonia; diagnostic; ultrasound; Pakistan; Mozambique
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Mozambique, cases
  Interventions: Device: Lung ultrasound
- Mozambique, controls
  Interventions: Device: Lung ultrasound
- Pakistan, cases
  Interventions: Device: Lung ultrasound
- Pakistan, controls
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound will be performed on all children to investigate imaging patterns characteristic of pneumonia.

SUMMARY:
The purpose of this study is to evaluate the impact of LUS on the diagnosis and management of childhood pneumonia in developing countries

ELIGIBILITY:
Inclusion Criteria (chest indrawing cases):

* Male or female, 2 through 23 months of age
* Cough <14 days or difficulty breathing
* Visible indrawing of the chest wall, with or without fast breathing
* Ability and willingness of child's caregiver to provide informed consent and to be available for follow-up for the planned duration of the study, including accepting a home visit if he/she fails to return to the study facility for a scheduled follow-up visit

Inclusion Criteria (non-chest indrawing controls):

* Male or female, 2 through 23 months of age
* Cough <14 days or difficulty breathing
* Ability and willingness of child's caregiver to provide informed consent and to be available for follow-up for the planned duration of the study, including accepting a home visit if he/she fails to return to the study facility for a scheduled follow-up visit

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cases will be children 2 through 23 months of age who present to a study hospital with history of cough or difficulty breathing and chest indrawing. Controls will be children 2 through 23 months of age who present with cough or difficulty breathing, but without chest indrawing, fast breathing or fever.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
LUS findings at enrollment | 8 hours

SECONDARY OUTCOMES:
Repeat LUS findings | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Centro de Investigação em Saúde de Manhiça (CISM), Manhiça, Mozambique
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Riaz A, Cambaco O, Ellington LE, Lenahan JL, Munguambe K, Mehmood U, Lamorte A, Qaisar S, Baloch B, Kanth N, Nisar MI, Volpicelli G, Bassat Q, Jehan F, Ginsburg AS. Feasibility, usability and acceptability of paediatric lung ultrasound among healthcare providers and caregivers for the diagnosis of childhood pneumonia in resource-constrained settings: a qualitative study. BMJ Open. 2021 Mar 11;11(3):e042547. doi: 10.1136/bmjopen-2020-042547. PMID 33707268
- [Derived] Lenahan JL, Volpicelli G, Lamorte A, Jehan F, Bassat Q, Ginsburg AS. Multicentre pilot study evaluation of lung ultrasound for the management of paediatric pneumonia in low-resource settings: a study protocol. BMJ Open Respir Res. 2018 Dec 19;5(1):e000340. doi: 10.1136/bmjresp-2018-000340. eCollection 2018. PMID 30622716